CLINICAL TRIAL: NCT02051699
Title: One-Leg Standing Radiograph: A Novel Technique to Evaluate the Severity of Knee Osteoarthritis
Brief Title: One-Leg Standing Radiograph: A Novel Technique to Evaluate the Severity of OA Knee
Acronym: OA knee
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Department of orthopeadic surgery, Thammasat University
Other Study IDs: orthoTU04
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Severity of OA Knee; Difference of Joint Space Width Between One-leg and Both-leg Standing Radiograph
Keywords: Osteoarthritis of the knee; Weight bearing radiograph; Kellgren-Lawrence classification; Joint space width; One-leg standing view
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- One-leg standing view
  Interventions: Procedure: radiographic of standing knee
- both-leg standing view
  Interventions: Procedure: radiographic of standing knee

INTERVENTIONS:
Procedure: radiographic of standing knee — the patients stand on their one leg with pillar support and both-leg then shoot the x-ray beam to their knee

SUMMARY:
The purpose of this study is assess the severity of osteoarthritic knee between one-leg and both-leg standing radiograph in primary OA knee

DETAILED DESCRIPTION:
All patients were performed digital radiographs which one-leg and both-leg standing anteroposterior view. Medial and lateral joint space width were measured. The severity of OA knee was identified by the Kellgren-Lawrence (KL) classification.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral knee pain more than 3 months

Exclusion Criteria:

* Inflammatory OA knee
* previous knee injury
* previous knee infection
* previous knee surgery
* pregnant women
* unable to bear weight on one leg

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who came to our clinic which bilateral knee pain
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change of joint space with between one-leg standing and both-leg standing radiographs in OA knee patients | one day

SECONDARY OUTCOMES:
Change of radiographic grading between one-leg and both-leg standing AP views in OA knee patients | one day

CONTACTS AND LOCATIONS:
Overall Officials: supakit kanitnate, M.D., Principal Investigator — orthopaedic department
Locations (1):
- department of orthopaedic surgery, Faculty of medicine, Thammasat university, Khlong Luang, Changwat Pathum Thani, Thailand